CLINICAL TRIAL: NCT04394039
Title: Effects of COVID-19-Related Self-isolation on Psychological Response to Different Outdoor Environments in Singapore - Before & After Brain and Behavior Study
Brief Title: Post-Pandemic Perception of Public Space in Singapore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Agnieszka Olszewska-Guizzo, Dr., National University of Singapore
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB_S-20-12
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Stress; Anxiety
Keywords: landscape; exposure; EEG; fNIRS; stress; urban; self-isolation; covid-19; pandemic; public space; brain
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: within-subjects before/ after study
Masking Description: participants do not know the hypothesis of the study, other people cannot influence the brainwave reaction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- public sp exposures (Experimental): All participants undergo the procedure of visiting all landscape exposures in a random order.
  Interventions: Other: Public space exposure

INTERVENTIONS:
Other: Public space exposure — landscapes with nature and/or classified as contemplative (through a CLM psychometric measure) are expected to elicit different brainwave oscillations as compared to noncontemplative ones.

SUMMARY:
In this study it is aimed to investigate the difference between the brain response to different urban environments in Singapore before and after the COVID-19 pandemic. The datasets acquired from 34 healthy individuals as part of ongoing study "Effects of Landscape on the Brain" (IRB Ref #: S-18-352) will be used. These datasets consist of neurophysiological data recordings and behavioral self-reported measures and were collected before 20 of January 2020. The same experimental protocol would be followed, given that the data collection in the lab-setting would start after 7 th May 2020/whenever research activities are allowed to resume, and the outdoor sessions after the "circuit-breaker" period in Singapore is over.

DETAILED DESCRIPTION:
The aim is to explore the difference between pre and post COVID-19-related isolation on their perception of green and public spaces, as well as mood, neuroelectrical (EEG) and haemodynamic (fNIRS) response.

The hypothesi is that crowded, busy public spaces, such as experimental site near Chinatown MRT, may induce more patterns of brain activity related to stress, anxiety and aversive attitudes after COVID-19 as compared to before. Similarily, it is expected that green urban spaces, such as experimental site at Hortpark, perceived after COVID-19 can elicit more salutogenic effect of relaxation, positive emotions and attention restoration than before the pandemic.

This study will allow better understanding of the mental health consequences of unprecedented period of isolation at home and social distancing. The relationship between city residents and their living environment may change due to COVID-19 and it's very important to uncover the mental health implications of social distancing to prepare for potential future outbreaks through developing tools and solutions addressing specific issues. Finally, for the urban planning and design the study may highlight important trends in changing human perception of space and redefine the concept of a "healthy city".

ELIGIBILITY:
Inclusion Criteria:

* Age of 21 to 75
* Right-handed only

Exclusion Criteria:

* left-handed
* serious visual or auditory impairment

  * Major neurological disorders e.g. epilepsy, stroke
  * Any form of cancer
  * Major heart diseases: e.g. ischemic heart disease
  * Major lung diseases: e.g. chronic obstructive pulmonary disorder.
  * Major liver disease e.g. liver failure
  * Major kidney disease e.g. kidney failure

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
EEG power in alpha band | 5 minutes
  predictor of positive affect and positive mental health outcomes, measured with EEG
EEG power in beta band | 5 minutes
  more beta in the right temporal lobes associated with stimuli-driven attention, measured with EEG
fNIRS haemodynamics | 5 minutes
  decreased oxy-hemoglobin in the frontal part of the brain indicates more relaxation

SECONDARY OUTCOMES:
Profile of mood states | 30 minutes
  self-reported, pre-and post- stimulation Profile of Mood States (POMS) scale measures the change in the momentary mood, giving as an outcome measure the Total Mood Disturbance (TMD), where 1 is neutral, and above 1 is disturbed mood
landscape preference measured with self-assessment manikin scale | 30 minutes
  measured using pictorial Self-Asessment Manikin (SAM) where score ranged from -3 to +3, where the lower the score the less positive (valence + arousal) emotions are caused by looking at the view

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Health Innovation & Technology (iHealthtech), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No